CLINICAL TRIAL: NCT06995040
Title: Initial Predictors of Long-term Brain Resilience After Minor Ischemic Stroke: a Study Nested in the Brest Stroke Population-based Registry
Brief Title: BREMISS : Brain Resilience Minor Stroke Study
Acronym: BREMISS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC23.0188 - BREMISS
Record Dates: First submitted 2025-05-21; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Stroke Ischemic
Keywords: stroke; Predictive model
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Retrospective study for pairing the population-based stroke registry and hospital medical record data and prospective study for calling back patient more than 4 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Minor ischemic stroke (Other): Patients registered in the Brest Stroke Registry who have been a minor stroke more than 4 years ago
  Interventions: Diagnostic Test: Cerebral MRI without contrast agent injection; Genetic: saliva sample; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: Cerebral MRI without contrast agent injection — Cerebral MRI at inclusion or after
Genetic: saliva sample — Saliva sample for DNA analysis at inclusion or send to their home.
Other: Questionnaires — Quality of life and cognitive questionnaires at inclusion

SUMMARY:
All patients eligible recorded in the Brest Stroke Registry (BSR) will be proposed to have either a telephone interview or a face-to-face interview.

In the case of telephone interview, they will be proposed to have a saliva kit for DNA analysis send to their home at the time as the self-questionnaires that will need to be send back to the hospital.

In the case of face-to-face interview, they will be proposed to have on the spot a saliva sample for DNA and a cerebral MRI.

Around 1000 patients can be included.

DETAILED DESCRIPTION:
The study is a retrospective study for pairing the population-based stroke registry and hospital medical record data and prospective study for calling back patient more than 4 years for new clinical, cognitive, thymic and quality of life evaluations and for DNA sample and cerebral MRI realization Duration of recruitment is anticipated to last between 2 years and 2 years and half.

The principal objective is to develop a predictive model of quality of life more than 4 years after stroke onset in patients with minor stroke based on initial (first days after stroke onset) patients characteristics based on the assumption that more than 4 years after a stroke the related sequelae are going to be stable.

ELIGIBILITY:
Inclusion Criteria:

* Cases of stroke in the Brest Stroke Registry (BSR)
* Ability to sign informed consent
* Patients followed-up > 4 years during the study period
* NIHSS score ≤ 5 on admission
* First stroke above 18 and before 75-year old
* Rankin before stroke < 1
* Possibility to draw saliva samples for genomic study
* Possibility to perform Cerebral MRI

Exclusion Criteria:

* Patients with transient neurological deficits resolving within one hour and normal brain imaging will be excluded.
* Not affiliated to social security
* Patient under legal protection or deprived of liberty by a judicial or administrative decision
* Patient unable to sign informed consent
* Patient whose follow-up will be impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life score | At inclusion
  Quality of life score is evaluated with the SF-36 questionnaire. It is a dichotomized score : good or bad recovery

SECONDARY OUTCOMES:
EQ5D score | At inclusion
  It is a questionnaire to describe patient's health with 5 items (Mobility; Autonomy; Activity; Pain/Discomfort; Anxiety/Depression) with 5 anwers each (No problem/light problems/moderate problem/serious problems/incapable)
Stroke Impact Scale | At inclusion
  Stroke Impact Scale includes 59 items and assesses 8 domains: Strength (4 items), Hand function (5 items), ADL/IADL (10 items), Mobility (9 items), Communication (7 items), Emotion (9 items), Memory and thinking (7 items), Participation/Role function (8 items)
Mortality | At inclusion
  Mortality is collected from the Brest Stroke Registry, and concerns patients who have been stroke 4 years ago.
Recurrence | At inclusion
  Recurrence is collected from the Brest Stroke Registry, and concerns patients who have been stroke 4 years ago.
Rankin score | At inclusion
  It is a scale about disability after stroke. The score is between 0 (no symptom) to 5 (serious disability). The study uses Rankin score dichotomized in good [0-1] and bad [2-5] prognosis.
Utility-Weighted Modified Rankin Scale | At inclusion
  The Modified Rankin Scale is a measure of functional outcome after stroke, evaluating the degree of disability or dependence in daily life. There is 7 grades ranging from 0 (no symptoms) to 6 (death).
WHO Disability Assessment Schedule (WHODAS) | At inclusion
  It is an auto-questionnaire of disability in daily life. There are 15 questions with 5 anwers ranging from 0 (No disability) to 5 (extreme disability/incapability)
Clinical Functioning Information Tool (ClinFIT) | At inclusion
  It is an auto-questionnaire to evaluate patient functioning. There are 30 questions, with score ranging from 0 (no problem) to 30 (complete problem).
Montreal Cognitive Assesment (MoCA) | At inclusion
  It is a cognition test with 7 items (visuospatial; designation; memory; attention; langage; abstraction; orientation). The total score is ranging from 0 to 30 points.
Mini Mental State Examination (MMSE) | At inclusion
  It is a cognition test with 6 items (orientation ; learning ; attention/calculation ; reminder; langage ; visuospatial constructive). The total score is ranging from 0 to 30 points.
Center for Epidemiologic Studies-Depression (CES-D) | At inclusion
  It is an auto-questionnaire to evaluate depression with 20 questions. There are 6 answers with score ranging from 0 to 6 (0 : Never/very rarely ; 1: rarely; 2 :quite often; 3: frequently/always).
Generalized Anxiety Disorder-7 (GAD-7) | At inclusion
  It is an auto-questionnaire for screening of generalized anxiety disorder with 7 questions. There are 4 answers : Never / Several days / More than half the days / Almost every day.
Primary Care PTSD Screen for DSM-5 (PTSD-5) | At inclusion
  It is an auto-questionnaire to evaluate stroke experience. there are 5 questions with 2 answers Yes/No
APATHY INVENTORY IA | At inclusion
  It is an auto-questionnaire to obtain information on the presence of apathy in patients with brain disorders. There are 3 items : emotional blunting; loss of initiative; loss of interest, with score ranging from 0 (mild) to 12 (severe).
Multidimensional Fatigue Inventory (MFI) | At inclusion
  It is an auto-questionnaire to evaluate fatigue. There are 10 items with score ranging from 1 (not agree at all) to 5 (completely agree)
Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) | At inclusion
  It is a questionnaire to evaluate cognitive declin, with 16 questions, with score ranging from 1 (much better) to 5 (much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Serge TIMSIT, Pr, Principal Investigator — CHU de Brest
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.